CLINICAL TRIAL: NCT03558841
Title: Effect of THERA-Trainer Lyra Gait Training in Addition to Physical Therapy on the Mobility of Geriatric Rehabilitation Inpatients Compared to Physical Therapy Alone: Randomized, Active-controlled, Parallel Group, Intervention Trial
Brief Title: Effect of Lyra Gait Training on the Mobility of Geriatric Rehabilitation Inpatients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment goal not met in allotted recruitment period
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC ID 2017-01495; SNCTP000002696 (Other: Swiss National Clinical Trials Portal (SNCTP))
Record Dates: First submitted 2018-05-16; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Mobility Limitation; Muscle Weakness
Keywords: gait; mobility; geriatric; rehabilitation; inpatient
MeSH Terms: conditions — Mobility Limitation; Muscle Weakness | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomized, active-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Gait training with the THERA-Trainer Lyra (3x/week) in addition to conventional geriatric rehabilitation physical therapy (6x/week) during inpatient period. After discharge home, continuation of Lyra gait training (3x/week), discontinuation of physical therapy.
  Interventions: Other: Gait training with the THERA-Trainer Lyra; Other: Physical therapy
- Control Group (Active Comparator): Conventional geriatric rehabilitation physical therapy (6x/week) during inpatient period. After discharge home, discontinuation of physical therapy.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Gait training with the THERA-Trainer Lyra — Gait training with the THERA-Trainer Lyra end-effector gait trainer 3x/week during the inpatient and the outpatient periods.
  Arms: Intervention Group
Other: Physical therapy — Conventional geriatric rehabilitation physical therapy (6x/week) during the inpatient period. After discharge home, discontinuation of physical therapy.

SUMMARY:
This study evaluates the effect of the addition of gait training to physical therapy on the gait of geriatric rehabilitation inpatients. Half of the patients will receive gait training with a gait training machine and conventional physical therapy in combination, the other half of the patients will receive conventional physical therapy alone.

DETAILED DESCRIPTION:
The geriatric rehabilitation inpatients recruited for this study primarily have difficulties with muscle weakness and walking generally due to a prolonged period of bed rest (as opposed to patients who primarily have cognitive disorders or neurological diseases), generalized muscle weakness and deconditioning. The rehabilitation goal for these patients is to be discharged home (not institutionalized) with improved mobility. Geriatric patients require intensive training in order to reach their pre-hospital levels of mobility and physical functional performance. Usual care involves physical therapy sessions, generally six times per week. Regaining mobility is crucial for quality of life and functional independence.

The aim of this intervention trial is to compare the effectiveness of Lyra gait training plus conventional physical therapy (intervention group) on gait compared to conventional physical therapy alone (control group) in geriatric rehabilitation patients. We hypothesize that, post-intervention, the intervention group will have better mobility and physical functional performance than the control group. Trial results will provide physical therapists and rehabilitation physicians with valuable information to better treat their inpatients and more efficiently use the limited time available for inpatient physical therapy sessions. Specifically, physical therapists should be better able to determine if the benefit of the Lyra gait trainer for geriatric rehabilitation inpatients with primarily muscle deconditioning is strong enough to warrant their extra time investment of providing the Lyra gait training. Results should also help determine in the future if the target population should continue with outpatient therapy after their discharge home. If this trial supports our hypothesis, then the trial results will provide data needed for the sample size calculation for a subsequent, larger trial.

The THERA-Trainer Lyra (from Ability AG, distributed by medica Medizintechnik GmbH) is an automated gait trainer with adjustable body weight support (no exoskeleton) and adjustable pedals (not a treadmill) that move in a physiological gait pattern derived from natural human walking movements. The upright position and the repetitive movement patterns activate muscle memory and allow safe gait training at the individual's performance limit throughout rehabilitation. The Lyra gait training is used to regain walking ability, improve gait speed, improve endurance and improve the gait pattern in geriatric rehabilitation patients.

Ten patients should be enrolled in this study:

Intervention group (n=5): Lyra gait training thrice weekly and conventional physical therapy (6 times per week) during inpatient period. After discharge home, continuation of thrice weekly Lyra gait training and discontinuation of physiotherapy.

Control group (n=5): Conventional physical therapy (6 times per week) during inpatient period. After discharge home, discontinuation of physical therapy.

At enrollment (Visit 1), all participants will be rehabilitation inpatients. The duration of the inpatient period will be determined clinically based on medical need and will thus vary from patient to patient. The average length of stay for the targeted population is approximately two weeks. Visit 2 will be performed shortly before the patient is discharged home. For each participant, the outpatient period (between Visit 2 and Visit 3) will be the same duration as the inpatient period (between Visit 1 and Visit 2).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Rehabilitation inpatients at Felix Platter Hospital with primarily muscle weakness and difficulty walking
* Community-dwellers before hospital admission with planned discharge home
* Body weight 150 kg or less
* Body height between 100 cm and 195 cm
* Mini-Mental State Examination score 21 points or more
* Signed informed consent for study participation

Exclusion Criteria:

* Clinically significant neurologic or musculoskeletal diseases which severly affect walking, e.g. advanced Parkinson's disease or hemiplegia
* Severe cardiac insufficiency
* Advanced chronic pulmonary disease (COPD Gold IV)
* Amputations of extremities (except missing fingers)
* Blindness
* Inability to understand and speak German well enough to understand the patient information, training and assessment instructions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Change in gait velocity | Baseline, after 2 weeks, after 4 weeks
  Habitual, preferred ("normal") walking speed (cm/s) quantified with the GAITRite electronic walkway system

SECONDARY OUTCOMES:
Change in grip strength | Baseline, after 2 weeks, after 4 weeks
  Grip strength (kg) of each hand (best result of two attempts for each hand used for data analysis)
Change in general mobility | Baseline, after 2 weeks, after 4 weeks
  Timed Up and Go Test time (seconds); faster test times represent better general mobility
Change in spatial-temporal gait parameters (other than walking velocity) | Baseline, after 2 weeks, after 4 weeks
  Gait parameters quantified with the GAITRite electronic walkway system
Change in endurance | Baseline, after 2 weeks, after 4 weeks
  Six Minute Walk Test; distance walked (meters) in six minutes; greater distance walked represents better endurance
Change in functionality (DEMMI total score, absolute values) | Baseline, after 2 weeks, after 4 weeks
  The de Morton Mobility Index (DEMMI) assesses functionality in different positions (lying, sitting, standing, walking); absolute values range from zero to 19 points; higher scores reflect better functionality
Change in functionality (DEMMI total score, scaled values) | Baseline, after 2 weeks, after 4 weeks
  The de Morton Mobility Index (DEMMI) assesses functionality in different positions (lying, sitting, standing, walking); scaled scores range from zero to 100 points; higher scores reflect better functionality
Change in fear of falling | Baseline, after 2 weeks, after 4 weeks
  Subjective fear of falling assessed by self-report using the "Falls Efficacy Scale-International Version (FES-I)" questionnaire; results range from 16 to 64 Points; higher scores reflect greater fear of falling; total number of points will be analysed
Change in subjective intensity of the Lyra training | Baseline, after 2 weeks, after 4 weeks
  Subjective intensity assessed by self-report using the "Borg Rating of Perceived Exertion Scale" questionnaire; score range from 6 (no exertion at all) to12 (maximal exertion); higher scores represent greater subjective intensity and exertion of the Intervention training
Change in the THERA-Trainer Lyra machine settings | Baseline, after 2 weeks, after 4 weeks
  Settings of the THERA-Trainer Lyra gait training machine

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A. Bridenbaugh, M.D, Principal Investigator — Head of the Basel Mobility Center of the Felix Platter Hospital
Locations (1):
- Felix Platter Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided